CLINICAL TRIAL: NCT07051083
Title: Intelligent Diagnosis of Bladder Cancer Staging and Prediction of New Adjuvant Chemotherapy Efficacy Based on Deep Learning and Transfer Learning in Ultrasound-Magnetic Resonance-Pathology Multimodal Multiscale
Brief Title: Bladder Cancer Staging and Prediction of New Adjuvant Chemotherapy Efficacy Based on Deep Learning and Transfer Learning in Ultrasound-Magnetic Resonance-Pathology Multimodal Multiscale
Acronym: MICS-BC
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Qiyun Ou, Dr., Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSKY-2023-1306-01; 2024A03J1194 (Other Grant/Funding Number: Guangzhou Science and Technology Bureau)
Record Dates: First submitted 2024-01-06; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Bladder Cancer; Staging; Deep Learning; Neoadjuvant Chemotherapy; Contrast Enhanced Ultrasound
Keywords: Bladder Cancer; Multi-omics; Staging; Deep Learning; Neoadjuvant Chemotherapy; Contrast Enhanced Ultrasound
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Training Group: Approximately 300 patients, which are used for the training dataset.
  Interventions: Diagnostic Test: Risk Stratification
- Internal Validation Group: Approximately 100 patients, which are used for internal validation to assess the accuracy of the model.
  Interventions: Diagnostic Test: Risk Stratification
- External Validation Group: Approximately 100 patients，which are used for external validation to assess the accuracy of the model.
  Interventions: Diagnostic Test: Risk Stratification

INTERVENTIONS:
Diagnostic Test: Risk Stratification — Risk Stratification for Assessing Muscle Infiltration in Bladder Cancer.

SUMMARY:
Bladder cancer is the most common malignant tumor of the urinary system. The presence or absence of muscle invasion in early bladder cancer is an independent prognostic factor. The involvement of muscle invasion affects the choice of surgical methods and treatment. Preoperatively, the precise assessment of bladder cancer staging has important practical value. A more accurate preoperative assessment of bladder cancer staging can reduce overtreatment and provide a favorable basis for clinicians to choose more reasonable and effective surgical methods. Clinically, there has been a longstanding desire to diagnose the staging of bladder cancer through a simple, convenient, effective, and non-invasive examination. As relevant research progresses, a multi-omics diagnostic model will be beneficial in improving diagnostic efficiency. This project aims to establish a multi-omics artificial intelligence system based on deep learning and transfer learning to accurately diagnose the staging of bladder cancer and predict the efficacy of neoadjuvant chemotherapy. This system will assist in clinical treatment decision-making.

DETAILED DESCRIPTION:
Research Content

1. Establishment of Ultrasound and Magnetic Resonance Imaging-Pathology-Clinical Dataset: This project aims to include medical records diagnosed through ultrasound and magnetic resonance imaging. Combining results from cytopathology or tissue pathology, the project will collect ultrasound images of the bladder, magnetic resonance images of the bladder, pathology images, and clinically relevant follow-up data. Tumor tissue specimens will be collected for immunohistochemical fluorescence staining. Participants with indistinct imaging findings or those with other primary malignant tumors will be excluded. The goal is to establish an ultrasound and magnetic resonance imaging-pathology-clinical dataset.
2. Establishment of an Artificial Intelligence System for Precise Diagnosis of Bladder Cancer Staging and Prognosis based on Ultrasound Imaging: Collecting clinical baseline information, surgical pathology, and ultrasound images of enrolled subjects. The ultrasound images will undergo homogenization processing. Utilizing algorithms based on U-Net, Transformer, and attention mechanisms for tissue segmentation and feature extraction, a deep learning model based on convolutional neural networks will be established for precise diagnosis of bladder cancer staging and prognosis:

   Construction of a mathematical model for staging bladder cancer using ultrasound contrast: Using convolutional neural networks for deep learning to build a mathematical model for staging bladder cancer. Developing an artificial intelligence diagnostic system for ultrasound contrast images based on deep learning and mathematical models to determine whether bladder cancer has muscle invasion.

   Construction of a mathematical model to discriminate prognosis features of bladder cancer using ultrasound imaging: Automatically delineating target areas and extracting ultrasound image features of bladder cancer lesions using new artificial intelligence technology - convolutional neural networks to build a model for evaluating the prognosis of bladder cancer lesions and achieving accurate prognosis diagnosis.
3. Establishment of an Artificial Intelligence System for the Joint Diagnosis of Bladder Cancer and Staging based on Ultrasound and Magnetic Resonance Imaging with Pathology: Based on bladder ultrasound, magnetic resonance imaging, and pathology image data, the baseline information of study subjects will be digitized. Ultrasound images, magnetic resonance images, and pathology images will undergo homogenization processing. Utilizing algorithms based on U-Net, Transformer, and attention mechanisms for segmentation and feature extraction of bladder ultrasound images, magnetic resonance images, and pathology images, a deep learning model based on convolutional neural networks will be established for the precise diagnosis of bladder cancer staging and prognosis:

   Construction of a mathematical model for joint pathology-based staging of bladder cancer using ultrasound and magnetic resonance imaging: Using convolutional neural networks for deep learning to build a mathematical model for staging bladder cancer. Based on the mathematical model, continuously optimizing algorithms, developing multi-omics, multidimensional artificial intelligence diagnostic systems based on ultrasound images, magnetic resonance images, pathology images, and clinical features, achieving accurate diagnosis of bladder cancer staging and prognosis prediction models.

   Construction of a mathematical model to discriminate prognosis features of bladder cancer using joint ultrasound, magnetic resonance, and pathology: Automatically delineating target areas and extracting features of bladder cancer lesions using convolutional neural networks and new artificial intelligence technology. Building a mathematical model to evaluate the prognosis of bladder cancer lesions.

   After the completion of the multi-omics, multidimensional artificial intelligence precise prediction model, validate the reliability of the model in prospective observational cohort study data and implement an intelligent system to assist in improving the efficiency of doctor diagnosis.
4. Establishment of an Artificial Intelligence System based on Dynamic Quantitative Immune Cell Maps using Ultrasound Imaging: Based on bladder ultrasound and pathological immunohistochemistry data, artificial intelligence algorithms will accurately determine the expression of immune cells through ultrasound images. Visualization of 2D spatial distribution heatmaps will be conducted to explore the intercorrelation features between ultrasound images and immune cells. Study subjects will be divided into training and validation cohorts. The baseline information of study subjects will be digitized. Ultrasound images will undergo homogenization processing. Utilizing algorithms based on U-Net, Transformer, attention mechanisms, and generative adversarial networks for tissue segmentation, feature extraction, and model establishment:

Construction of a mathematical model for quantitative immune cell maps using ultrasound images: Using new artificial intelligence technology - convolutional neural networks for deep learning to build a mathematical model for predicting the expression of immune cells. Developing an artificial intelligence diagnostic system for quantifying the microenvironment of ultrasound contrast images, determining the expression of immune cells in bladder cancer lesions.

The model will combine the immune cells with the 2D ultrasound image prediction heatmap, forming a visual 2D ultrasound image-immune cell heatmap. Exploring the spatial location of immune cells in ultrasound images. Using single-cell and spatial transcriptome sequencing methods to verify the accuracy of the spatial distribution of ultrasound image-quantified immune cells.

ELIGIBILITY:
Inclusion Criteria:

1. Ultrasound and other imaging examinations (CT, MR, etc.) suggest bladder masses and are suspicious for bladder cancer patients.
2. The bladder is well filled, and no allergic reactions to ultrasound contrast agents are found.
3. No surgery or radiotherapy/chemotherapy has been performed.
4. Patients who meet the indications for surgical resection and are planned for surgical treatment, including one of the following:

   1. Clinical symptoms consistent with suspected bladder cancer (such as gross hematuria, etc.);
   2. Patients with confirmed primary or recurrent bladder cancer by cystoscopic biopsy;
   3. Rapid urine cytology and urine cytology FISH testing suggest malignancy.

Exclusion Criteria:

1. Individuals unable to tolerate surgery;
2. Individuals allergic to ultrasound contrast agents, unable to undergo ultrasound contrast examination;
3. Unsuccessful preoperative ultrasound contrast examination or non-compliant patients;
4. Postoperative pathology does not indicate bladder cancer;
5. Patients who have undergone chemotherapy or radiation therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 480 patients who were diagnosed with bladder cancer based on postoperative pathology at Sun Yat-sen Memorial Hospital, Sun Yat-sen University will be included between January 2023 and December 2026.
Sampling Method: Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of Muscle Invasion in Bladder Cancer | Perform contrast-enhanced ultrasound (CEUS) examination within 2 weeks before the procedure.
  To evaluate the preoperative staging of bladder cancer，whether it is non-muscle invasive bladder cancer (NMIBC) or muscle invasive bladder cancers (MIBC)

SECONDARY OUTCOMES:
Evaluate the Diagnostic Performance of Deep Learning and Transfer Learning in Preoperative Prediction of Muscle-Invasive Status in Bladder Cancer | The patient should return for follow-up at 3 months postoperatively
  The diagnostic performance of the Deep Learning and Transfer Learning Model was primarily evaluated using the statistical metrics of AUC (Area Under the ROC Curve), sensitivity, specificity, accuracy, negative predictive value (NPV), and positive predictive value (PPV).

CONTACTS AND LOCATIONS:
Overall Officials: Qiyun Ou, Dr., Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP, Analytic Code

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Antoni S, Ferlay J, Soerjomataram I, Znaor A, Jemal A, Bray F. Bladder Cancer Incidence and Mortality: A Global Overview and Recent Trends. Eur Urol. 2017 Jan;71(1):96-108. doi: 10.1016/j.eururo.2016.06.010. Epub 2016 Jun 28. PMID 27370177
- [Background] Humphrey PA, Moch H, Cubilla AL, Ulbright TM, Reuter VE. The 2016 WHO Classification of Tumours of the Urinary System and Male Genital Organs-Part B: Prostate and Bladder Tumours. Eur Urol. 2016 Jul;70(1):106-119. doi: 10.1016/j.eururo.2016.02.028. Epub 2016 Mar 17. PMID 26996659
- [Background] Flaig TW, Spiess PE, Agarwal N, Bangs R, Boorjian SA, Buyyounouski MK, Chang S, Downs TM, Efstathiou JA, Friedlander T, Greenberg RE, Guru KA, Guzzo T, Herr HW, Hoffman-Censits J, Hoimes C, Inman BA, Jimbo M, Kader AK, Lele SM, Michalski J, Montgomery JS, Nandagopal L, Pagliaro LC, Pal SK, Patterson A, Plimack ER, Pohar KS, Preston MA, Sexton WJ, Siefker-Radtke AO, Tward J, Wright JL, Gurski LA, Johnson-Chilla A. Bladder Cancer, Version 3.2020, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2020 Mar;18(3):329-354. doi: 10.6004/jnccn.2020.0011. PMID 32135513
- [Background] Grossman HB, Natale RB, Tangen CM, Speights VO, Vogelzang NJ, Trump DL, deVere White RW, Sarosdy MF, Wood DP Jr, Raghavan D, Crawford ED. Neoadjuvant chemotherapy plus cystectomy compared with cystectomy alone for locally advanced bladder cancer. N Engl J Med. 2003 Aug 28;349(9):859-66. doi: 10.1056/NEJMoa022148. PMID 12944571
- [Background] Yin M, Joshi M, Meijer RP, Glantz M, Holder S, Harvey HA, Kaag M, Fransen van de Putte EE, Horenblas S, Drabick JJ. Neoadjuvant Chemotherapy for Muscle-Invasive Bladder Cancer: A Systematic Review and Two-Step Meta-Analysis. Oncologist. 2016 Jun;21(6):708-15. doi: 10.1634/theoncologist.2015-0440. Epub 2016 Apr 6. PMID 27053504
- [Background] Winquist E, Kirchner TS, Segal R, Chin J, Lukka H; Genitourinary Cancer Disease Site Group, Cancer Care Ontario Program in Evidence-based Care Practice Guidelines Initiative. Neoadjuvant chemotherapy for transitional cell carcinoma of the bladder: a systematic review and meta-analysis. J Urol. 2004 Feb;171(2 Pt 1):561-9. doi: 10.1097/01.ju.0000090967.08622.33. PMID 14713760
- [Background] Seiler R, Ashab HAD, Erho N, van Rhijn BWG, Winters B, Douglas J, Van Kessel KE, Fransen van de Putte EE, Sommerlad M, Wang NQ, Choeurng V, Gibb EA, Palmer-Aronsten B, Lam LL, Buerki C, Davicioni E, Sjodahl G, Kardos J, Hoadley KA, Lerner SP, McConkey DJ, Choi W, Kim WY, Kiss B, Thalmann GN, Todenhofer T, Crabb SJ, North S, Zwarthoff EC, Boormans JL, Wright J, Dall'Era M, van der Heijden MS, Black PC. Impact of Molecular Subtypes in Muscle-invasive Bladder Cancer on Predicting Response and Survival after Neoadjuvant Chemotherapy. Eur Urol. 2017 Oct;72(4):544-554. doi: 10.1016/j.eururo.2017.03.030. Epub 2017 Apr 5. PMID 28390739
- [Background] Makboul M, Farghaly S, Abdelkawi IF. Multiparametric MRI in differentiation between muscle invasive and non-muscle invasive urinary bladder cancer with vesical imaging reporting and data system (VI-RADS) application. Br J Radiol. 2019 Dec;92(1104):20190401. doi: 10.1259/bjr.20190401. Epub 2019 Oct 8. PMID 31573328
- [Background] Sidhu PS, Cantisani V, Dietrich CF, Gilja OH, Saftoiu A, Bartels E, Bertolotto M, Calliada F, Clevert DA, Cosgrove D, Deganello A, D'Onofrio M, Drudi FM, Freeman S, Harvey C, Jenssen C, Jung EM, Klauser AS, Lassau N, Meloni MF, Leen E, Nicolau C, Nolsoe C, Piscaglia F, Prada F, Prosch H, Radzina M, Savelli L, Weskott HP, Wijkstra H. The EFSUMB Guidelines and Recommendations for the Clinical Practice of Contrast-Enhanced Ultrasound (CEUS) in Non-Hepatic Applications: Update 2017 (Long Version). Ultraschall Med. 2018 Apr;39(2):e2-e44. doi: 10.1055/a-0586-1107. Epub 2018 Mar 6. PMID 29510439
- [Background] Hu FB. Metabolic profiling of diabetes: from black-box epidemiology to systems epidemiology. Clin Chem. 2011 Sep;57(9):1224-6. doi: 10.1373/clinchem.2011.167056. No abstract available. PMID 21690202
- [Background] Ou Q, Yu Y, Li A, Chen J, Yu T, Xu X, Xie X, Chen Y, Lin D, Zeng Q, Zhang Y, Tang X, Yao H, Luo B. Association of survival and genomic mutation signature with immunotherapy in patients with hepatocellular carcinoma. Ann Transl Med. 2020 Mar;8(5):230. doi: 10.21037/atm.2020.01.32. PMID 32309377
- [Background] Yu Y, Zeng D, Ou Q, Liu S, Li A, Chen Y, Lin D, Gao Q, Zhou H, Liao W, Yao H. Association of Survival and Immune-Related Biomarkers With Immunotherapy in Patients With Non-Small Cell Lung Cancer: A Meta-analysis and Individual Patient-Level Analysis. JAMA Netw Open. 2019 Jul 3;2(7):e196879. doi: 10.1001/jamanetworkopen.2019.6879. PMID 31290993